CLINICAL TRIAL: NCT00581854
Title: Phase II Pilot Study of Hyper-CVAD Plus Rituximab for Previously Untreated Mantle Cell Lymphoma
Brief Title: Phase 2 Hyper-CVAD/Rituximab for Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO00401
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-06

CONDITIONS: Mantle Cell Lymphoma
Keywords: untreated mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: modified Hyper-CVAD — rituximab and modified hyperfractionated cyclophosphamide, vincristine doxorubicin, dexamethasone (hyperCVAD) administered every 28 days for 4-6 cycles followed by rituximab maintenance therapy consisting of four weekly doses every six months for two years

SUMMARY:
rituximab and modified (hyperCVAD) administered every 28 days for 4-6 cycles followed by rituximab maintenance therapy consisting of four weekly doses every six months for two years

DETAILED DESCRIPTION:
rituximab and modified hyperfractionated cyclophosphamide, vincristine doxorubicin, dexamethasone (hyperCVAD) administered every 28 days for 4-6 cycles followed by rituximab maintenance therapy consisting of four weekly doses every six months for two years

ELIGIBILITY:
Inclusion Criteria:

* Untreated mantle cell lymphoma

Exclusion Criteria:

* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-06; Primary Completion 2006-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad S Kahl, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UWCCC, Madison, Wisconsin, United States

REFERENCES:
- [Result] Kahl BS, Longo WL, Eickhoff JC, Zehnder J, Jones C, Blank J, McFarland T, Bottner W, Rezazedeh H, Werndli J, Bailey HH; Wisconsin Oncology Network. Maintenance rituximab following induction chemoimmunotherapy may prolong progression-free survival in mantle cell lymphoma: a pilot study from the Wisconsin Oncology Network. Ann Oncol. 2006 Sep;17(9):1418-23. doi: 10.1093/annonc/mdl127. Epub 2006 Jun 9. PMID 16766582

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Single Arm Maintenance rituximab following induction chemoimmunotherapy
Period: Overall Study
Arm/Group | Rituximab
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: SAEs during induction therapy
Arm/Group | Group 1
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate to Induction Therapy
Description: Outcome is the % of subjects who achieved a Complete Response (CR) or Complete Response Unconfirmed (CRu) after induction therapy, following the Cheson et al criteria for standardized response criteria (1999).
Time Frame: Median follow up of 37 months
Population: All Subjects enrolled were included in the analysis. Response rate is represented as % of total subjects enrolled.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Group 1: All subjects received R-HyperCVAD induction therapy.
Arm/Group | Group 1
Number analyzed (Participants) | 22
percentage of participants | 64 [44 to 80]

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 8/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=22)
Infection with febrile neutropenia, Gr 3 (Infections and infestations) | 2 (2)
Neutropenic Fever Gr 3 (Blood and lymphatic system disorders) | 4 (4)
Atrial fibrillation gr 3, dyspnea (Cardiac disorders) | 1 (1)
perionitis, gr 5 (Infections and infestations) | 1 (1) — bowel infarction resulting in septicemia
psuedomonas sepsis, gr 5 (Infections and infestations) | 1 (1)
Hyponatremia, gr 3 (Metabolism and nutrition disorders) | 1 (1)
Chronic Heart Failure, gr 5 (Cardiac disorders) | 1 (1) — Pt also experienced sinus tachycardia, hypotension.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=22)
Neutropenia (Blood and lymphatic system disorders) | 18 (59) — 19 events of gr 3, 41 events of Gr 4 = 59 events out of 104 cycles of therapy adminsitered.
febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) — Events are total occurrences out of 104 cycles of therapy adminsitered across subjects
infection with neutropenia (Infections and infestations) | 6 (6) — total is # of grade 3 and 4 events in 104 cycles of therapy administered across 22 subjects.
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (24) — 22 cases of grade 3, 2 cases of gr 4 thrombocytopenia out of 104 cycles of therapy administered.
Anemia (Blood and lymphatic system disorders) | 8 (12) — 11 cases of grade 3, 1 case of gr 4 anemia out of 104 cycles of therapy administered.
Hyperglycemia (Metabolism and nutrition disorders) | 4 (9) — 9 cases of gr 3 hyperglycemia out of 104 cycles of therapy administered.
dehydration (General disorders) | 1 (3) — 3 cases of gr 3 dehydration out of 104 cycles of therapy administered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes